# **Informed consent form**

| Title of research programme: Clinical study on the prevention |
|-------------------------------------------------------------------------|
| and treatment of postoperative metastasis in stage IIA-IIIA lung cancer |
| with negative expression of driver genes by Fuzheng Quxie Recipe |
| Research organization: Shanghai Municipal Hospital of |
| Traditional Chinese Medicine |
| Principal Investigator: Jianhui Tian |
| Vargian No. 1.0, 2022 12.21 |
| Version No.: 1.0, 2022.12.21 |

# **Informed Consent Form • Informed Communication**

# **Page**

Dear patient: you as a patient after radical lung adenocarcinoma with clinical stage IIA-IIIA

#### Dear Sir/Madam:

We would like to invite you to take part in a clinical study of "Clinical study on the prevention and treatment of postoperative metastasis of stage IIA-IIIA lung cancer with negative expression of driver genes by Fuzheng Quxie Formula".

Before you decide whether or not to participate in this study, please read the following as carefully as possible.

#### 1. Introduction of the study

As the most common malignant tumour of the respiratory system, primary bronchopulmonary cancer has a high mortality rate perennially ranking first among all kinds of malignant tumours, which greatly threatens the life and health of human beings. In China, the latest data show that there are about 787,000 new cases of lung cancer, with an incidence rate of 57.26/100,000, which ranks the first in the national morbidity and cause of death of all genders. Therefore, metastasis of lung cancer after radical treatment is a difficult problem limiting the improvement of the overall efficacy of the treatment, and at the same time, the cost of treatment caused by metastasis of the lung cancer has caused great economic pressure on the society and families. At the same time, the treatment cost caused by postoperative metastasis has also caused enormous economic pressure on society and families.

The current standard treatment after radical lung cancer treatment is mainly chemotherapy, but the clinical benefit is limited. Guided by the academic thought of "treating cancer by reforcing healthy qi" and based on the theory of "Deficiency of Vital Qi and Hidden Toxin", Fuzheng Quxie Formula has gained a high level of evidence of preventing the recurrence and metastasis of early stage lung cancer after surgery, and revealing the mechanism of its regulation of immune system to prevent and control the metastasis.

Based on the theory of "Deficiency of Vital Qi and Hidden Toxin", this project will conduct a high level multi-centre clinical study of Chinese and Western medicine to prevent and treat patients with kinesin-negative lung adenocarcinoma after radical surgery. By designing a rigorous randomised controlled clinical trial and adopting the standard postoperative adjuvant therapy and Fuzheng Quxie Formula, the applicant will confirm the effectiveness and safety of TCM in preventing and treating metastasis of Stage IIA-IIIA lung adenocarcinoma patients with negative expression of kinesiology, and provide high-level evidence-based medical evidence of TCM in preventing and treating metastasis of Stage IIA-IIIA lung adenocarcinoma patients with negative expression of kinesiology. To develop TCM diagnostic and treatment protocols and guidelines for TCM intervention in postoperative metastasis of stage IIA-IIIA lung adenocarcinoma with negative driver gene expression. At the same time, we will clarify the clinical characteristics of the immune system, circulating tumour cells and MRD expression of patients with driver gene expression-negative stage IIA-IIIA lung adenocarcinoma, explore the predictive indexes of the efficacy of driver gene expression-negative stage IIA-IIIA lung adenocarcinoma, and establish the predictive model of the efficacy of treatment; we will also elucidate the targets of TCM in preventing postoperative metastasis of driver gene expression-negative stage IIA-IIIA lung adenocarcinoma, and explain the mechanism of supporting the positive and dispelling the evil. We will explain the targets of Chinese medicine in preventing postoperative metastasis of stage IIA-IIIA lung adenocarcinoma with negative expression of driver genes and the mechanism of "Deficiency of Vital Qi", so as to provide the basis for entering the relevant guidelines.

During the course of the study, you will be asked to 1) complete the entire course of treatment (a total of 32 treatments) as scheduled by the researcher; 2) fill out questionnaires and answer questions from the researcher to evaluate the efficacy of the treatment programme during the study (a total of 7 times, before treatment, at weeks 4, 8 and 12, and at the end of the entire course of treatment at months 1, 3, and 6, respectively), and we ask for your support. Support.

Your participation in this study is completely voluntary, and you may withdraw from the study at any time during the treatment period without affecting your relationship with your doctor or causing you to suffer any loss of medical or other benefits, and you will continue to be seen effectively by your doctor in the normal course of medical treatment.

The study will be conducted in accordance with the principles of (the Declaration of Helsinki) and your right to privacy will be strictly protected. All information from the study will be kept strictly confidential and your private information will not be included in the study summary report or in the published literature. The study has been ethically reviewed by the Medical Ethics Committee and has

been deemed safe and ethical, and the research has been conducted in strict compliance with the spirit of  $\langle$  the Declaration of Helsinki $\rangle$ .

#### 2. Inclusion and exclusion criteria

#### 2.1 Inclusion criteria:

- 2.1.1 Patients with clinical stage IIA-IIIA lung adenocarcinoma after radical surgery, patients within 6 weeks after surgery;
- 2.1.2 Driver gene negative (no EGFR, ALK, ROS1 mutation), PD-1/L1 expression <1%;
- 2.1.3 Meet the diagnostic criteria for the lung qi and yin deficiency type, with primary symptoms of cough, low sputum volume, shortness of breath, low or muted voice, weakness, and thirst without desire to drink. Secondary symptoms include spontaneous sweating, nocturnal sweating, five heartburns, red tongue or teeth marks on the edge of the tongue, and weak pulse. At least two primary symptoms and one of the secondary symptoms are present;
- 2.1.4 Patients aged between 18 and 75 years;
- 2.1.5 Patients with basically normal blood routine and biochemical indexes, etc., without serious viral or bacterial infections; patients without organ failure and serious heart disease (blood bilirubin <68  $\mu$ mol/L, aspartate aminotransferase <90 IU/L, creatinine <350  $\mu$ mol/L, leukocyte count >3.5×109/L and less than 12×109/L, platelet count >80×109/L, erythrocyte pressure area >0.20);
- 2.1.6 Those with a tumour PS score of ≤2 and no other serious comorbidities;
- 2.1.7 I gave informed consent to participate in the study, signed the informed consent form and had good compliance;
- 2.1.8 Non-pregnant and lactating patients;
- 2.1.9 Chemotherapy-related indicators are qualified;
- 2.1.10 Those who have no allergic reaction to the ingredients in the formula.

## 2.2 Exclusion criteria (including suspension criteria)

- 2.2.1 Patients who are incompletely resected or whose cancer has undergone recurrence or metastasis;
- 2.2.2 Patients who are being treated with other drugs or therapeutic methods (including other Chinese herbal medicines, immunological drugs, radiotherapy, etc.);
- 2.2.3 Patients who are themselves mentally ill and have a lack of autonomous behaviour;
- 2.2.4 Women who are pregnant, preparing for pregnancy or breastfeeding;
- 2.2.5 Patients with combined serious diseases of heart, lung, brain, liver, kidney and haematopoietic system, and psychiatric patients;
- 2.2.6 People with allergies or known hypersensitivity to the components of this drug;
- 2.2.7 Patients who are participating in other clinical trials or have participated in other clinical trials within 3 months;
- 2.2.8 Alcoholism and/or psychoactive substances, drug abusers and dependent persons;
- 2.2.9 other pathologies or conditions that, in the judgement of the investigator, have the effect of reducing the likelihood of enrolment or complicating enrolment, e.g. frequent changes in the work environment, unstable living conditions, etc., that predispose to loss of visits.

# 3 What will I need to do if I take part in the study?

- 3.1 Before you are enrolled in the study, you will undergo the following tests to determine if you are ready to take part in the study, and your doctor will ask about, and record, your physical examination of you.
- 3.2 We will tell you truthfully that you have an equal chance of being placed in the treatment group and the control group, and that if you agree and are eligible for enrolment, the researcher will arrange for you to be placed in both the treatment group and the control group, based on random sampling. Patients participating in this study will have an equal chance of being assigned to both groups and will be entered into the study after meeting the NAC criteria. Standardised postoperative adjuvant treatment will be given to both the treatment and control groups, and an assessment of your condition will be carried out after your treatment.
- 3.3 Other Matters Requiring Your Cooperation: You must follow the doctor's instructions to carry out the treatment on time, and please promptly and objectively reflect to the doctor the changes in your condition after each treatment, and fill in the scoresheet for evaluation on time. If you have other medical conditions that require you to continue taking medication, please inform your doctor. If you need other treatment during the study, please contact your doctor in advance. Stay comfortable and as emotionally stable as possible during treatment. You will need to come to our clinic for treatment and follow-up visits, as well as physical, chemical, and immunological tests and imaging tests, which may be inconvenient for you during the study.

# 4. Benefits of participating in the study

You and the community may benefit from this study. Such benefits include the possibility that your condition and quality of life may improve, and that this study may provide good guidance for clinical treatment and better use of TCM in tumour patients, but it cannot be ruled out that this study will not improve your condition.

## 5. Risks of participating in research

The unit responsible for the study will make every effort to prevent and treat any harm that may occur as a result of this study. If during the study you experience any discomfort, a new change in your condition, or any unforeseen circumstances, whether or not related to the treatment, you should notify your doctor promptly and we will make a judgement and medical treatment. During the trial, there may be adverse reactions to the medication, such as nausea and vomiting, stomach upset and some other discomforts, so please tell your study physician immediately and he/she will deal with any discomfort you experience.

A professional oncologist will be in charge of this trial. If you experience any discomfort during the use of the drug, including dizziness, nausea, loss of appetite, drowsiness, constipation and itching of the skin, etc., please contact the researchers in the study group immediately, and we will provide you with a reasonable, safe and effective solution.

During the study period, you will be required to visit our clinic on time for treatment and follow-up, and to have some physicochemical and immunological tests and imaging tests, which may cause you trouble or inconvenience.

## 6. Compensation for participation in the study

We will provide you with herbal treatment during the treatment period and give each subject who cooperates in the participation and completion of the trial a travelling allowance of \$100 at the end of the treatment.

# 7. Is personal information confidential?

Your medical records (study chart/CRF, physical and chemical examination reports, etc.) will be kept intact at the hospital. The investigator, sponsor's representative, and ethics committee will be allowed to access your medical records. Any public reports about this study will not disclose your personal identity. Every effort will be made to protect the privacy of your personal medical information to the extent permitted by law.

#### 8. How can I get more information?

You may ask any questions about this study at any time.

Your doctor will give you his/her phone number so that he/she can answer your questions.

Your doctor will keep you informed if there is any important new information during the study that may affect your willingness to continue participating in the study.

# 9. Voluntary Options for Participation and Withdrawal from the Study

Whether or not you participate in this study is entirely up to you. You may refuse to take part in this study, or you may leave the study at any time during the study. If you choose to leave this study, your benefits will not be affected and you will not be discriminated against or retaliated against for doing so. Your participation in this study may be discontinued at any time by your doctor or the researcher in the best interest of you.

If you withdraw from the study for any reason, you may be counselled about your use of the study drug. You may also be asked to undergo laboratory tests and a physical examination if your doctor deems it necessary. You may also refuse and will not be discriminated against or retaliated against for doing so.

If you choose to participate in this study, we expect you to stay for the full duration of the study.

If you do not participate in this study, or if you withdraw from the study, there are many alternatives such as exercise therapy, cognitive-behavioural therapy, psychological interventions, and so on. You do not have to choose to participate in this study in order to treat your disease.

If you do choose to take part in this study, we hope that you will stay with us for the full duration of the study.

# 10. What should I do now?

It is up to you to decide whether or not you want to participate in this study. You can discuss your decision with your family or friends.

Please ask your doctor as many questions as possible before you make your decision to take part in the study until you fully understand the study.

## 11. Ethics Committee

If you have questions or need to ask someone other than the investigator, please consult the Ethics Committee of Shanghai Hospital of Traditional Chinese Medicine.

Ethics Committee Office: 2nd Floor, Building 9, Shanghai Hospital of Traditional Chinese Medicine, Shanghai, China.

**Tel:** 56628310

Thank you for reading the above material. If you decide to take part in this study, please let your doctor know and he/she will organise everything for you regarding the study.

Please keep this material with you

# **Informed Consent** • Consent Signature Page

**Project name:** Clinical study of Fuzheng Expectorant Formula against postoperative metastasis of stage IIA-IIIA lung cancer with negative expression of driver gene

Version number: V1.0

Version Date: 21 Feb 2023

#### **Statement of Consent:**

I have read the above description of this study and have had the opportunity to discuss and ask questions about this study with my doctor.

All the questions I have asked have been answered to my satisfaction.

I am aware of the possible risks and benefits of participating in this study. I understand that participation in the study is voluntary and I confirm that I have had sufficient time to think about it and understand it:

I can ask my doctor for more information at any time.

I can withdraw from this study at any time without discrimination or retaliation, and that my medical treatment and rights will not be affected.

I am equally aware that if I withdraw from the study, it would be in my own best interests and that of the study as a whole if I informed my doctor of any changes in my condition and completed the appropriate physical and physical-chemical examinations.

If I take any other medication due to the needs of my illness, I will seek my doctor's advice beforehand or tell him/her truthfully afterwards.

I give my consent to the doctors of the Oncology Department of the Shanghai Hospital of Traditional Chinese Medicine, representatives of the Ethics Committee and other departments to have access to my study materials.

I will be provided with a signed and dated copy of the informed consent form.

| Finally, I have decided to agree | to participate in | this study and | promise to | follow my |
|---|---|---|---|---|
| doctor's instructions as much as | possible. | | | |

| Subject's signature: | Date: | Month | Day |
|--------------------------------------|-------|-------|-----|
| Subject's contact telephone number:_ | | | |

| I confirm that I have explained to the subject the details of thi his/her rights and possible benefits and risks, and given him/her a informed consent form. | • |
|---|---|
| Signature of the investigator:Date:Year | Month |
| Investigator contact phone number: | |